CLINICAL TRIAL: NCT00761969
Title: Prevention of Ischemic Events in Patients With Peripheral Arterial Disease by the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice
Brief Title: Prevention of Ischemic Events in Patients With Peripheral Arterial Disease
Acronym: PID-PAB
Status: Completed | Type: Observational
Sponsor: KRKA (Industry)
Collaborators: University Medical Centre Ljubljana (Other); University of Ljubljana School of Medicine, Slovenia (Other); Krka, d.d., Novo mesto, Slovenia (Unknown)
Responsible Party: Sponsor
Other Study IDs: PID-PAB
Record Dates: First submitted 2008-09-28; First posted 2008-09-30 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; secondary prevention; cardiovascular /atherothrombotic events; European guidelines; Cardiovascular disease prevention
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood (16 ml) for analysis of inflammatory markers (from serum) and genotyping, to be correlated with clinical outcomes.
  Anonymity of patients is proveded by coding the samples and the patients clinical records.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PAB: Subjects with stable peripheral arterial disease; ankle-brachial pressure index on at least one leg =< 0.90.
  Interventions: Other: Implementation of the European Guidelines on cardiovascular Disease Prevention in Clinical Practice
- Control: Subjects without peripheral arterial disease (palpable pedal pulses and a normal ankle-brachial pressure index of 0.91-1.30), age- and sex-matched to the stuy group with PAD
  Interventions: Other: Implementation of the European Guidelines on cardiovascular Disease Prevention in Clinical Practice

INTERVENTIONS:
Other: Implementation of the European Guidelines on cardiovascular Disease Prevention in Clinical Practice — Life-style modification advice and prescribing standard cardioprotective medication (antiplatelet agents, statins, antihypertensive agents) according to the European Guidelines on Cardiovascular Disease Prevention in Clinical practice.

SUMMARY:
The PID-PAB study aims to test the efficacy of the European Guidelines on Cardiovascular Disease Prevention in patients with peripheral arterial disease. Survival, the rate of major atherothrombotic events (myocardial infarction, stroke, critical limb ischemia) and the incidence of revascularization procedures will be compared between a group of patients with stable peripheral arterial disease (PAD) and age- and sex-matched control subjects without PAD. Both groups will be receiving up-to-date medical care according to their cardiovascular risk based on the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice. Yearly follow-up is planned for 5 years. The PID PAB study aims to test (a) whether stable PAD is still an adverse prognostic indicator in spite of contemporary preventive measures, and (b) to what extent do contemporary preventive measures improve the prognosis of patients with PAD in comparison to historic controls, representing the natural history of the disease.

DETAILED DESCRIPTION:
The observational study Prevention of Ischemic Events in Patients with Peripheral Arterial Disease by the European Guidelines on Cardiovascular Disease Prevention (Slovenian acronym of the study: PID-PAB)aims to test the efficacy of the European Guidelines on Cardiovascular Disease Prevention in patients with peripheral arterial disease, who have an even higher mortality rate than patients with isolated coronary artery disease or cerebrovascular disease when left to the natural course of the disease. The PID-PAB study will compare the rates of survival, major atherothrombotic events (myocardial infarction, stroke, critical limb ischemia) and revascularization procedures between a group of patients with stable peripheral arterial disease (PAD) and a control group of age- and sex-matched subjects without PAD. Both groups will be receiving up-to-date medical care (including life-style advice and prescription of cardioprotective medication) according their cardiovascular risk based on the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice. PAB is defined by a reduced ankle-brachial pressure index of =< 0.90, while absence of PAD is defined by palpable pedal pulses and a normal ankle-brachial index (0.91-1.30). Exclusion criteria are: age < 40 or > 80 years at inclusion, active cancer or other disease with a life expectancy of les than 5 years, any major atherothrombotic event in 30 days prior to enrollment, and pregnancy. All subjects will be followed annually for 5 years by comprehensive medical examinations. The settings of the study are primary care facilities in Slovenia, European Union. The target size of each group is 1000 subjects, i.e., 5000 patient years. The number of participating physicians-researchers is estimated at 100, with a goal for each physician to recruit 10 patients with PAD and 10 age- and sex-matched controls. The study is coordinated by a steering committee consisting of researchers from the Department of Vascular Diseases at the University of Ljubljana Medical Centre, Institute of Biomedical Informatics at the University of Ljubljana School of Medicine, Department of Family Medicine at the University of Ljubljana School of Medicine and the pharmaceutical company Krka, Slovenia, who is also the sponsor of the study. The protocol of the study has been approved by the Committee of Medical Ethics of the Republic of Slovenia.

The PID PAB study aims to answer the questions:

1. Is stable PAD is still an adverse prognostic indicator in spite of contemporary preventive measures?
2. To what extent do contemporary preventive measures improve the prognosis of patients with PAD in comparison to historic controls (described in earlier reports on the natural history of PAD ? We expect to still find a significant difference in the rate of cardiovascular events between patients with PAD and their peers without PAD, but we hypothesize that contemporary preventive measures will strongly attenuate the adverse prognosis of PAD regarding survival and major atherothrombotic events in comparison to the natural history of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PAD: ankle-brachial pressure index <= 0.90
2. Controls: palpable pedal pulses, ankle-brachial pressure index 0.91-1.30

Exclusion Criteria:

1. Age < 40 or > 80 years at inclusion
2. Malignancy with a life expectancy < 5 years
3. Atherothrombotic event within a month before inclusion (acute coronary syndrome, stroke or documented transient ischemic attack, critical limb ischemia)
4. pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stable, objectively confirmed PAD, recruited from primary care settings in Slovenia, Europe.
  Control subjects of comparable age- and sex-distribution, without PAD, recruited from primary care settings in Slovenia, Europe.
Sampling Method: Non-Probability Sample
Enrollment: 1455 (Actual)
Dates: Start 2004-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ales Blinc, MD, DSc, Principal Investigator — Dept of Vascular Diseases, University of Ljubljana Med Ctr
Locations (1):
- Department of Vascular Diseases, University of Ljubljana Medical Center, Ljubljana, Slovenia

REFERENCES:
- [Background] Criqui MH, Langer RD, Fronek A, Feigelson HS, Klauber MR, McCann TJ, Browner D. Mortality over a period of 10 years in patients with peripheral arterial disease. N Engl J Med. 1992 Feb 6;326(6):381-6. doi: 10.1056/NEJM199202063260605. PMID 1729621
- [Background] Newman AB, Shemanski L, Manolio TA, Cushman M, Mittelmark M, Polak JF, Powe NR, Siscovick D. Ankle-arm index as a predictor of cardiovascular disease and mortality in the Cardiovascular Health Study. The Cardiovascular Health Study Group. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):538-45. doi: 10.1161/01.atv.19.3.538. PMID 10073955
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Background] De Backer G, Ambrosioni E, Borch-Johnsen K, Brotons C, Cifkova R, Dallongeville J, Ebrahim S, Faergeman O, Graham I, Mancia G, Manger Cats V, Orth-Gomer K, Perk J, Pyorala K, Rodicio JL, Sans S, Sansoy V, Sechtem U, Silber S, Thomsen T, Wood D; Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. European guidelines on cardiovascular disease prevention in clinical practice. Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. Eur Heart J. 2003 Sep;24(17):1601-10. doi: 10.1016/s0195-668x(03)00347-6. No abstract available. PMID 12964575
- [Background] Giampaoli S, Capewell S, Shelley E, Allender S, Briggs A, Jorgensen T, Labarthe D, Marques-Vidal P, Stegmayr B, Verschuren WM, Zdrojewski T. Foreword. Eur J Cardiovasc Prev Rehabil. 2007 Dec;14 Suppl 3:S1. doi: 10.1097/01.hjr.0000296928.40040.b0. No abstract available. PMID 18091132
- [Derived] Blinc A, Kozak M, Sabovic M, Bozic Mijovski M, Stegnar M, Poredos P, Kravos A, Barbic-Zagar B, Stare J, Pohar Perme M. Survival and event-free survival of patients with peripheral arterial disease undergoing prevention of cardiovascular disease. Int Angiol. 2017 Jun;36(3):216-227. doi: 10.23736/S0392-9590.16.03731-7. Epub 2016 Jun 22. PMID 27332992
- [Derived] Blinc A, Kozak M, Sabovic M, Bozic M, Stegnar M, Poredos P, Kravos A, Barbic-Zagar B, Pohar Perme M, Stare J; PID-PAB Investigators. Prevention of ischemic events in patients with peripheral arterial disease design, baseline characteristics and 2-year results an observational study. Int Angiol. 2011 Dec;30(6):555-66. PMID 22233617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 85 primary care physicians-researchers from Slovenia, acountry with a population of about 2 million. Participating physicians were educated on cardiovascular disease prevention according to the European guidelines attended annual progress report meetings and were visited at least once a year by a study monitor.
  .
Groups:
- Peripheral Arterial Disease: Subjects with stable peripheral arterial disease; ankle-brachial pressure index on at least one leg =< 0.90.
  Implementation of the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice: Life-style modification advice and prescribing standard cardioprotective medication (antiplatelet agents, statins, antihypertensive agents) according to the European Guidelines on Cardiovascular Disease Prevention in Clinical practice .
- Control: Subjects without peripheral arterial disease (palpable pedal pulses and a normal ankle-brachial pressure index of 0.91-1.30), age- and sex-matched to the stuy group with PAD
  Implementation of the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice: Life-style modification advice and prescribing standard cardioprotective medication (antiplatelet agents, statins, antihypertensive agents) according to the European Guidelines on Cardiovascular Disease Prevention in Clinical practice .
Period: Overall Study
Arm/Group | Peripheral Arterial Disease | Control
Started | 742 | 713
Completed | 542 | 573
Not Completed | 200 | 140
Not completed — Death | 112 | 47
Not completed — Lost to Follow-up | 88 | 93

BASELINE CHARACTERISTICS:
Groups:
- Peripheral Arterial Disease: Subjects with stable peripheral arterial disease; ankle-brachial pressure index on at least one leg =< 0.90.
  Implementation of the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice: Life-style modification advice and prescribing standard cardioprotective medication (antiplatelet agents, statins, antihypertensive agents) according to the European Guidelines on Cardiovascular Disease Prevention in Clinical practice (Eur Heart J 2003; 24: 1601-10, Eur J Cardiovasc Prev Rehabil. 2007;14 Suppl 2:S1-113).
- Control: Subjects without peripheral arterial disease (palpable pedal pulses and a normal ankle-brachial pressure index of 0.91-1.30), age- and sex-matched to the stuy group with PAD
  Implementation of the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice: Life-style modification advice and prescribing standard cardioprotective medication (antiplatelet agents, statins, antihypertensive agents) according to the European Guidelines on Cardiovascular Disease Prevention in Clinical practice (Eur Heart J 2003; 24: 1601-10, Eur J Cardiovasc Prev Rehabil. 2007;14 Suppl 2:S1-113).
- Total: Total of all reporting groups
Arm/Group | Peripheral Arterial Disease | Control | Total
Number analyzed (Participants) | 742 | 713 | 1455
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.8) | 64.7 (9.2) | 64.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 275 | 552
  Male | 465 | 438 | 903
Region of Enrollment [Number; unit: participants]
  Slovenia | 742 | 713 | 1455

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Major Cardiovascular Events
Description: Total number of deaths, cardiovascular deaths, non-fatal myocardial infarctions, ischemic strokes and critical limb ischemia.
Time Frame: 5 years:
Measure: Number; unit: participants
Arm/Group | Peripheral Arterial Disease | Control
Number analyzed (Participants) | 742 | 713
participants
  Death of all causes | 112 | 47
  Cardiovascular death | 51 | 17
  Non-fatal myocardial infarction | 50 | 21
  Non-fatal ischemic stroke | 22 | 14
  Critical limb ischemia | 11 | 0
Statistical Analysis 1: Comparison: Peripheral Arterial Disease vs Control; Survival, major-event-free survival and event-free survival of patients with PAD and control subjects was estimated by the Kaplan-Meier method and compared by the log-rank test. The numbers of non-fatal events and revascularization procedures (which could be more than one per person) were compared using the Poisson regression - the outcome being the number of events per person-year; Test type: Superiority or Other; p < 0.001, Log Rank

2. Secondary Outcome: Incidence of Revascularization Procedures
Description: Incidence of coronary, carotid and peripheral arterial revascularization procedures
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Peripheral Arterial Disease | Control
Number analyzed (Participants) | 742 | 713
participants
  Peripheral arterial revascularization | 183 | 2
  Coronary revascularization | 64 | 20
  carotid revascularization | 31 | 8
  Abdominal aortic revascularization | 6 | 0

ADVERSE EVENTS:
Time Frame: Death of all causes, non-fatal major ischemic events (myocardial infarction, ischemic stroke, critical limb ischemia) and revascularization procedures were recorded yearly for 5 years.
Description: At the time of yearly follow-up, non-fatal major ischemic events and revascularization procedures in the previous year were recorded according to medical records. In case of a "no show" on a scheduled visit, subjects or their relatives and their family physician were actively contacted.
Arm/Group | Peripheral Arterial Disease | Control
Serious Adverse Events (participants affected / at risk) | 195/742 | 82/713
Other Adverse Events (participants affected / at risk) | 284/742 | 30/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Arterial Disease (N=742) | Control (N=713)
Death of all causes (General disorders) | 112 (112) | 47 (47)
Non-fatal myocardial infarction (Cardiac disorders) | 50 (50) | 21 (21)
Non-fatal ischemic stroke (Nervous system disorders) | 22 (22) | 14 (14)
Critical limb ischemia (Vascular disorders) | 11 (11) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Arterial Disease (N=742) | Control (N=713)
Peripheral arterial revascularization procedure (Vascular disorders) | 183 (183) | 2 (2) — Endovascular or surgical peripheral arterial revascularization
Coronary revascularization procedure (Vascular disorders) | 64 (64) | 20 (20) — Percutaneous coronary intervention or surgical coronary revascularization
Carotid revascularization (Vascular disorders) | 31 (31) | 8 (8) — Surgical carotid endarterectomy or carotid artery stenting
Abdominal aortic revascularization (Vascular disorders) | 6 (6) | 0 (0) — Surgical aortic repair or endovascular aortic repair (EVAR)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No